CLINICAL TRIAL: NCT06924268
Title: Evaluating the Impact of a Single Art Therapy Session on Mood and Symptom Burden in Palliative Care Patients
Brief Title: Impact of a Single Art Therapy Session on Mood and Symptom Burden in Palliative Care
Status: Not yet recruiting | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025060172580
Record Dates: First submitted 2025-03-31; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Emotional Distress; Pain; Anxiety
Keywords: Palliative; End of life; art therapy; quality of life
MeSH Terms: conditions — Pain; Anxiety Disorders; Death

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Single Art Therapy Session — Each participant will engage in a 30-60 minute structured art therapy session using pre-drawn coloring sheets featuring themes such as mandalas, nature scenes, and inspirational designs. A variety of coloring tools will be provided, including crayons, colored pencils, markers, gel pens, and watercolor paints. Sessions will be facilitated by the primary investigator, who will provide non-directive prompts and engage in casual conversation to foster comfort and engagement.
  Other Names: Visual arts therapy; Expressive arts

SUMMARY:
The goal of this observational study is to explore whether a single art therapy session can improve mood and reduce symptom burden in adult palliative care patients at a Canadian inpatient unit. The main questions it aims to answer are:

* Does a single art therapy session reduce overall symptom burden, as measured by the Edmonton Symptom Assessment System (ESAS)?
* Does a single art therapy session improve mood, as measured by the Positive and Negative Affect Schedule (PANAS)?

Participants will:

* Complete two short questionnaires (ESAS and PANAS) before and after the session
* Participate in a 30-60 minute individual art therapy session

DETAILED DESCRIPTION:
This is a single-centre, prospective, observational pre-post study conducted at the QEII Health Sciences Centre, VG, 7A Palliative Care Unit. The aim is to evaluate whether a one-time, individualized art therapy session can positively impact emotional well-being and symptom distress in adults receiving inpatient palliative care.

Participants will be approached by the charge nurse and invited to participate if they meet the eligibility criteria. Following informed consent, participants will complete two validated self-report tools: the Edmonton Symptom Assessment System (ESAS) and the Positive and Negative Affect Schedule (PANAS). These assessments will be administered immediately before and again immediately after a 30-60 minute art therapy session, which will include open-ended creative engagement using simple materials such as watercolor and pastels.

The Study Objectives are:

1. To determine whether participation in a structured art therapy session improves mood and symptom burden in palliative care patients
2. Examine whether engagement in coloring activities influences emotional well-being as measured by the Positive and Negative Affect Schedule (PANAS) and symptom burden as measured by the Modified Edmonton Symptom Assessment System (ESAS).
3. Is there a difference in as-needed (PRN) opioid, benzodiazepine, and Z drug use in the 48 hours before and after the session
4. Examine whether specific patient characteristics, such as primary diagnosis or time from admission to intervention, impact the observed effects.

All data will be de-identified and analyzed descriptively and inferentially to assess trends in mood and symptom change following the intervention. This study does not involve randomization or a control group. It is designed to inform future research and program development in supportive care interventions within palliative settings.

ELIGIBILITY:
Inclusion Criteria:

* inclusion if they are adults (=18 years old)
* admitted to the PCU
* have the ability to communicate
* complete self-assessments with or without facilitator assistance
* possess the ability to engage in a 30-60 minute art therapy session

Exclusion Criteria:

* Patients will be excluded if they are under 18 years of age
* within 48hrs of admission or discharge
* experiencing severe cognitive impairment, uncontrolled symptoms, or delirium.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Palliative Care In-Patients at the VG, 7A Palliative Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Scores Measured by PANAS Before and After Art Therapy | Immediately before and immediately after the art therapy session
  The Positive and Negative Affect Schedule (PANAS) will be administered immediately before and immediately after a single art therapy session. PANAS is a self-reported 20-item scale measuring two mood domains: positive affect (10 items) and negative affect (10 items). Each item is rated on a scale from 1 (very slightly or not at all) to 5 (extremely), with subscale scores ranging from 10 to 50. Higher positive affect scores indicate more positive mood; higher negative affect scores indicate more distress.
Change in Symptom Burden Measured by Modified ESAS Before and After Art Therapy | Immediately before and immediately after the art therapy session
  The Edmonton Symptom Assessment System (ESAS) will be used to assess physical and emotional symptom burden immediately before and immediately after the art therapy session. ESAS consists of 9 core symptoms (e.g., pain, fatigue, nausea, anxiety, depression) each rated on a numeric scale from 0 (none) to 10 (worst possible severity). A total symptom score is calculated as the sum of all items, with higher scores indicating greater symptom burden. We will be using a modified version that does not include nausea, drowsiness, loss of appetite and dyspnea. The symptom "sadness" will be added to our assessment.

SECONDARY OUTCOMES:
Changes in PRN Opioid Use in the 48 Hours Before and After Art Therapy | 48 hours before and 48 hours after the art therapy session
  The total dosage (mg), number of doses, medication type, and route of administration of PRN opioid medications (e.g., hydromorphone, morphine) will be extracted from the medical chart for each participant for the 48 hours before and the 48 hours after the art therapy session. Data will be converted to oral morphine equivalents as applicable. Data will be analyzed to assess changes in frequency or total daily dose following the intervention.
Changes in PRN Benzodiazepine and Z-Drug Use in the 48 Hours Before and After Art Therapy | 48 hours before and 48 hours after the art therapy session
  The total dosage (mg), number of doses, medication type, and route of administration of PRN benzodiazepines (e.g., lorazepam) and Z-drugs (e.g., zopiclone) will be recorded from participant medical charts for the 48 hours before and after the art therapy session. Data will be analyzed to assess changes in frequency or total daily dose following the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Lees, MA, MSc, MD, FRCPC, Study Chair — Nova Scotia Health Authority; Jonathan Clements, BSc, Principal Investigator — Dalhousie University; Lindsay Flinn, MD, CCFP (PC), Study Chair — Nova Scotia Health Authority

IPD SHARING:
Plan to Share IPD: No